CLINICAL TRIAL: NCT06863610
Title: Investigating the Knee Extension Deficit on Knee Strength Recovery Following an Anterior Cruciate Ligament Reconstruction
Brief Title: Knee Extension Deficit Following an Anterior Cruciate Ligament Reconstruction (Extension Loss)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Leyla Eraslan, Associate Professor, Hacettepe University
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/140
Record Dates: First submitted 2025-02-22; First posted 2025-03-07 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Anterior Cruciate Ligament Injuries
Keywords: ACL; reconstruction; knee; extension deficit
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Extension Deficit (>5 degrees) (Experimental): Patients who had a knee extension ROM deficit of more than 5 degrees in the fourth week will be subject to the rehabilitation program under the supervision of the same physiotherapist 3 days a week for a period of 12 weeks. The rehabilitation program will include cold therapy, electrotherapy, and exercises focusing on improving knee functioning and restoring muscle strength. From 12 weeks to 6 months, a home exercise program will be advised to all patients equally.
  Interventions: Other: Extension Deficit (>5 degrees)
- Extension Deficit (<5 degrees) (Active Comparator): Patients who had a knee extension ROM deficit of less than 5 degrees in the fourth week will be subject to the rehabilitation program under the supervision of the same physiotherapist 3 days a week for a period of 12 weeks. The rehabilitation program will include cold therapy, electrotherapy, and exercises focusing on improving knee functioning and restoring muscle strength. From 12 weeks to 6 months, a home exercise program will be advised to all patients equally.
  Interventions: Other: Extension Deficit (<5 degrees)

INTERVENTIONS:
Other: Extension Deficit (>5 degrees) — Patients who had a knee extension ROM deficit of more than 5 degrees will included
  Arms: Extension Deficit (>5 degrees)
Other: Extension Deficit (<5 degrees) — Patients who had a knee extension ROM deficit of less than 5 degrees will included
  Arms: Extension Deficit (<5 degrees)

SUMMARY:
Knee extension loss following an anterior cruciate ligament (ACL) reconstruction is believed to play an important role in quadriceps strength recovery. One of the main goals of the rehabilitation following ACL reconstruction is to restore knee extensor muscle strength. Deficits of more than a five-degree extension range of motion (ROM) could lead to delayed knee functionality and anterior knee pain. However, the effect of knee extension deficits in the early postoperative phase of the ACL reconstruction on knee extensor muscle strength recovery and knee functionality is not yet known.

This study aimed to investigate the difference between knee extensor muscle strength recovery and knee functionality in patients with ACL repair who had a knee extension ROM deficit (>5°) in the early postoperative period and those who did not.

DETAILED DESCRIPTION:
Knee range of motion deficits are significant surgical complications following an anterior cruciate ligament (ACL) reconstruction, and despite current advances in surgical techniques, knee range of motion cannot always be regained. Previous studies reported that knee range of motion (ROM) deficits play an important role in knee extensor muscle weakness and knee osteoarthritis. Thus, deficits in knee extension joint motion are more difficult to tolerate than flexion deficits. It has been reported that a five-degree decrease in the extension ROM of the affected knee compared to the healthy side can lead to secondary complications such as difficulty walking and anterior knee pain. However, the effect of knee extension deficits in the early postoperative phase of the ACL reconstruction on knee extensor muscle strength recovery and knee functionality is not yet known.

This study aimed to investigate the difference between knee extensor muscle strength recovery and knee functionality in patients with ACL repair who had a knee extension ROM deficit (>5°) in the early postoperative period and those who did not.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent ACL repair using hamstring tendon autograft
* volunteered to participate in the study between the ages of 18-45
* a non-contact injury mechanism
* a Tegner Activity Score >5 before the injury
* regularly attended the rehabilitation program after surgery (not missing more than three sessions)

Exclusion Criteria:

* Patients who underwent ACL repair with patellar tendon autograft or allograft, revision surgery
* underwent meniscus and or cartilage repair in addition to ACL repair
* a history of previous knee, ankle, or groin injuries
* concomitant systemic and/or neurological pathologies
* a history of injury to the contralateral lower extremity
* do not want to participate in the evaluations that should be done before the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-15 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Quadriceps Muscle Strength Recovery | Qudriceps muscle strength will be measured at 4th weeks (isometric), 12 th weeks (isometric and concentric), 6th months (isometric, concentric, and eccentric) following a surgery.
  Isometric, concentric and eccentric quadriceps muscle strength will be measured using an isokinetic dynamometer (IsoMed®2000 D&R GmbH, Germany).
Hamstring Muscle Strength Recovery | Hamstring muscle strength will be measured at 4th weeks (isometric), 12 th weeks (isometric and concentric), 6th months (isometric, concentric, and eccentric) following a surgery.
  Isometric, concentric and eccentric hamstring muscle strength will be measured using an isokinetic dynamometer (IsoMed®2000 D&R GmbH, Germany).

SECONDARY OUTCOMES:
The Y Balance Test. Functional Testing 1 | Assessments will be conducted at 12th weeks and 6th months following a surgery
  The Y Balance Test will be used. Three repetitions will be conducted for each limb, and mean values were recorded in centimeters.
The Vertical Jump Test. Functional Testing 2 | Assessments will be conducted at 12th weeks and 6th months following a surgery
  The Vertical Jump Test will be used. Three repetitions will be conducted for each limb, and mean values were recorded in centimeters.
The Single Leg Hop Test. Functional Testing 3 | Assessments will be conducted at 12th weeks and 6th months following a surgery
  The Single Leg Hop Test will be used. Three repetitions will be conducted for each limb, and mean values were recorded in centimeters
The Lysholm score. Patient-reported outcomes measures 1 | Self-reported recovery will be recorded at 12th weeks and 6th months following a surgery
  The Lysholm score will be used to assess self-reported recovery. The Lysholm score is an eight-item questionnaire that evaluates patients following knee ligament injury. This is scored on a 100-point scale from 0 (worst symptoms) to 100 (best symptoms), with 25 points attributed to pain, 15 to locking, 10 to swelling, 25 to instability,10 to stair climbing and 5 points each to limping, use of a support and squatting.
The International Knee Documentation Committee subjective knee form (IKDC). Patient-reported outcomes measures 2 | Self-reported recovery will be recorded at 12th weeks and 6th months following a surgery
  The International Knee Documentation Committee subjective knee form (IKDC) will be used to assess self-reported recovery.
  IKDC subjective knee form contains 18 selected items designed to measure symptoms. Total IKDC score ranges from 0 to 100, with 100 indicating the absence of symptoms and higher levels of knee function.

CONTACTS AND LOCATIONS:
Overall Officials: Leyla Eraslan, Ph. D., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)